CLINICAL TRIAL: NCT04690595
Title: A Phase 1 Study Evaluating BAFFR-targeting CAR T Cells for Patients With Relapsed or Refractory B-cell Acute Lymphoblastic Leukemia
Brief Title: BAFFR Targeting CAR-T Cells for the Treatment of Relapsed or Refractory B-cell ALL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PeproMene Bio, Inc. (Industry)
Collaborators: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMB-101
Record Dates: First submitted 2020-12-24; First posted 2020-12-30 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Relapsed or Refractory B-cell Acute Lymphoblastic Leukemia
Keywords: B cell; ALL; relapsed or refractory
MeSH Terms: conditions — Recurrence; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BAFFR-CAR T cells (Experimental): B-cell activating factor receptor-Chimeric antigen receptor T cells
  Interventions: Biological: BAFFR-CAR T cells

INTERVENTIONS:
Biological: BAFFR-CAR T cells — First-in-human trial examining the safety and preliminary efficacy of BAFFR-CAR T cells in participants with r/r B-ALL

SUMMARY:
A Phase 1 Study Evaluating BAFFR-targeting CAR T Cells for Patients with Relapsed or Refractory B-cell Acute Lymphoblastic Leukemia

DETAILED DESCRIPTION:
This phase I trial evaluates the side effects and best dose of BAFFR-CAR T cells in treating patients with B-cell Acute Lymphoblastic Leukemia that has come back (recurrent) or does not respond to treatment (refractory). T cells are infection fighting blood cells that can kill cancer cells. The T cells given in this study will come from the patient and will have a new gene put in them that makes them able to recognize BAFFR, a protein on the surface of cancer cells. These BAFFR-specific T cells may help the body's immune system identify and kill BAFFR+ cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Documented informed consent of the participant and/or legally authorized representative.
2. Agreement to allow the use of archival tissue from diagnostic tumor biopsies. If unavailable, exceptions may be granted with study PI approval.
3. Age ≥ 18 years.
4. ECOG ≤ 2.
5. Life expectancy ≥ 16 weeks.
6. Histologically confirmed B-ALL or B-cell lymphoblastic lymphoma
7. Relapsed/refractory disease after failure of ≥ 2 prior lines of therapy.
8. Evidence of active BAFF-R expression at the time of enrollment.
9. Recovered to ≤ Grade 1 from the acute toxic effects (except alopecia) of prior anti-cancer therapy.
10. No known contraindications to leukapheresis, steroids or tocilizumab.
11. Ineligible for or failed prior CD19-targeted immunotherapy (e.g., blinatumomab or CD19-CAR T cells).

    For participants who had prior CD19-CAR T cell therapy:

    - At least 90-days has elapsed since participant received last CD19-CAR T cell therapy.

    AND

    - Persistence of prior CD19-CAR T cells must be evaluated and found to be <5% prior to leukapheresis procedure
12. Participants with CNS involvement by leukemia (CNS2 and asymptomatic CNS3) may be considered eligible after discussions with the study team.
13. Total serum bilirubin ≤ULN (unless has Gilbert's disease, then ≤3.0)
14. AST ≤ ULN
15. ALT ≤ ULN
16. Creatinine clearance of ≥ 40 mL/min per 24-hour urine test or the Cockcroft-Gault formula
17. Left ventricular ejection fraction (LVEF) ≥ 50%
18. O2 saturation ≥ 92% on room air.
19. Seronegative for HIV Ag/Ab combo, HCV*, and active HBV (Surface Antigen Negative)

    *If positive, Hepatitis C RNA quantitation must be performed and must be undetectable.
20. Women of childbearing potential (WOCBP): negative urine or serum pregnancy test If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
21. QuantiFERON-TB Gold or equivalent*

    *Results do not impact patient eligibility, however the test must be initiated prior to enrollment
22. Agreement by females and males of childbearing potential^ to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy.

    ^Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).
23. A complete liver evaluation (which includes ultrasound elastography, MRI of the liver and a hepatology consult) may be done if needed based on PI's recommendation.
24. Evaluation of acquired hemochromatosis (indicated through MRI of the liver and elevated levels of Ferritin) is recommended for participants who have undergone multiple transfusions and prior alloHCT.

Exclusion Criteria:

1. Autologous/allogeneic stem cell transplant within 100 days at the time of enrollment.
2. Immunosuppressant medications within 1 months prior to protocol enrollment.
3. Concurrent use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of inhaled steroids is not exclusionary. Physiologic replacement of steroids (prednisone ≤ 7.5 mg /day or equivalent) is allowed
4. Auto-immune disease or active GVHD within 4 months prior to protocol enrollment requiring systemic immunosuppressant therapy.
5. Class III/IV cardiovascular disability according to the New York Heart Association (NYHA) Classification.
6. Subjects with clinically significant arrhythmia or arrhythmias not stable on medical management within 2 weeks of enrollment.
7. Any abnormal liver enzyme levels (as defined ≥ULN in ALT, AST, Bilirubin and Alkaline Phosphatase levels) at time of enrollment
8. . Subjects with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system, including seizure disorder.
9. History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent.
10. Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia.
11. History of venous occlusive disease (VOD), or GvHD.

    a. Subjects with a history of the following GvHD may still be included in the study: i. Resolved Grade 2 or less steroid-sensitive acute skin GvHD ii. Grade 1 gastro-intestinal (GI)-GvHD developed within 100 days post prior alloHCT.

    iii. Limited chronic GvHD
12. History of stroke or intracranial hemorrhage within 6 months of enrollment.
13. History of other malignancies, except for malignancy surgically resected (or treated with other modalities) with curative intent, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; non-muscle invasive bladder cancer; malignancy treated with curative intent with no known active disease present for ≥ 3 years.
14. Clinically significant uncontrolled illness.
15. Active systemic uncontrolled infection requiring antibiotics.
16. Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection.
17. Females only: Pregnant or breastfeeding.
18. Any other condition that would, in the investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns with clinical study procedures.
19. Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-05-18 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2027-11-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 1 year post treatment
  Toxicity will be graded per Common Terminology Criteria for Adverse Events version 5.0, Cytokine Release Syndrome (CRS) and neurotoxicity which use the American Society for Transplantation and Cellular Therapy Consensus Criteria (ASTCT) and Graft versus Host Disease (GVHD) criteria. Toxicities will be followed from the start of lymphodepletion until the end of the study.

SECONDARY OUTCOMES:
Disease response | Up to 1 year post treatment
  Defined as complete response [CR], or complete response with incomplete blood count recovery [CRi], or complete response with partial hematological recovery [CRh]. Response will be evaluated using European Leukemia Net (ELN) criteria. Rates and associated 95% binomial exact confidence limits will be estimated (CR/CRi/CRh) rate.
Minimal residual disease (MRD) | Up to 1 year post treatment
  Negative MRD is defined by malignant cells < 0.01% by flow cytometry or clonoSEQ.
B cell frequency | Up to 1 year post treatment
  Measured by serum IgG level
Severity of graft-versus-host disease (GVHD) in recipients of prior allogeneic hematopoietic stem cell transplantation | Up to 1 year post treatment.
  Defined per Keystone criteria for acute GVHD and revised National Institute of Health (NIH) consensus on grading of chronic GVHD.
Progression-free survival (PFS) | From T cell infusion to the first observation of disease relapse/progression or death from any cause, whichever occurs first, assessed up to 15 years.
  Kaplan-Meier product limit method with log-log transformation for the confidence interval will be used to estimate PFS.
Overall survival (OS) | From the day of BAFFR-CAR T cell infusion to death from any cause assessed, up to 15 years.
  Kaplan-Meier product limit method with log-log transformation for the confidence interval will be used to estimate OS.

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Aldoss, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No